CLINICAL TRIAL: NCT02344875
Title: Clinical Pharmacological Study of FYU-981 Administered to Male and Female Elder or Non-elder Subjects
Brief Title: Clinical Pharmacology of FYU-981 (Elder Subjects)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-004
Record Dates: First submitted 2015-01-18; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — dotinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Male elder subjects (Experimental): Male 65- Years
  Interventions: Drug: FYU-981, (Oral single dosing)
- Male non-elder subjects (Experimental): Male 20-35 Years
  Interventions: Drug: FYU-981, (Oral single dosing)
- Female elder subjects (Experimental): Female 65- Years
  Interventions: Drug: FYU-981, (Oral single dosing)
- Female non-elder subjects (Experimental): Female 20-35 Years
  Interventions: Drug: FYU-981, (Oral single dosing)

INTERVENTIONS:
Drug: FYU-981, (Oral single dosing)

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety and pharmacodynamics after single oral administration of FYU-981 to male and female elder subjects in comparison with non-elder subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adult subjects
* 20-35 Years (non-elder groups)
* 65- Years (elder groups)
* Body mass index: >=18.5 and <25.0

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 48 hours
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 48 hours
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 48 hours
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 48 hours
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (kel: Elimination rate constant) | 48 hours
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed | 48 hours
Pharmacokinetics (MRT: Mean residence time) | 48 hours
Pharmacokinetics (Ae: Amount of drug excreted in urine) | 48 hours
Pharmacokinetics (fe: Fraction of dose excreted in urine) | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Tokyo, Japan

REFERENCES:
- [Derived] Nakatani H, Fushimi M, Sasaki T, Okui D, Ohashi T. Clinical pharmacological study of dotinurad administered to male and female elderly or young subjects. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):8-16. doi: 10.1007/s10157-019-01836-0. Epub 2019 Dec 30. PMID 31889230